CLINICAL TRIAL: NCT05893173
Title: Pilot Study: Establishing Glutamatergic Changes as the Mechanism of Action in the Rapid Antidepressant Effects of Sleep Deprivation
Brief Title: Pilot Study: Establishing Glutamatergic Changes in Rapid Antidepressant Effects of Sleep Deprivation
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 853162
Record Dates: First submitted 2023-05-12; First posted 2023-06-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Major Depressive Disorder: Ten individuals (aged 18-85) with a DSM-V diagnosis of MDD will undergo baseline GluCEST imaging and waking EEG prior to and following approximately 30 hours of total sleep deprivation.
  Interventions: Behavioral: Sleep Deprivation

INTERVENTIONS:
Behavioral: Sleep Deprivation — Ten individuals (aged 18-85) with a DSM-V diagnosis of MDD will undergo baseline GluCEST imaging prior to and following approximately 30 hours of total sleep deprivation.

SUMMARY:
In the treatment of Major Depressive Disorder (MDD), total sleep deprivation can produce rapid but short-lasting improvements in mood. In order to develop a new generation of treatments with rapid and sustained efficacy, a better understanding of the mechanism of action is urgently needed. One candidate mechanism is the modulation of synaptic strength mediated by glutamatergic activity as sleep deprivation has been suggested to increase synaptic strength. Although determining how sleep deprivation impacts the glutamatergic system is essential to isolating its mechanism of action, the invasive nature of most assessment methods has limited our ability to do so in humans. The proposed research aims to determine if changes in glutamatergic activity, reflecting the modulation of synaptic strength, underlie the antidepressant effects of sleep deprivation. In this project, the investigators will utilize a novel measure of glutamate imaging, GluCEST, to assess changes in glutamatergic activity, in addition to using a proxy measure, waking EEG theta activity, to assess synaptic strength following total sleep deprivation. Ten individuals (aged 18-85) with a DSM-V diagnosis of MDD will undergo baseline GluCEST imaging and waking EEG prior to and following approximately 30 hours of total sleep deprivation. Both clinician-administered and subjective mood measures will be collected. It is predicted that sleep deprivation will improve mood and increase glutamatergic activity and synaptic strength. Results from this project have the potential to identify the modifiable mechanisms by which rapid antidepressants work which could ultimately stimulate the development of novel interventions that work through the modulation of glutamatergic activity.

DETAILED DESCRIPTION:
Consent and Virtual Screening Participants who meet initial inclusion criteria via phone screen will be invited to the complete a virtual visit that will include additional screening (e.g. Medical history), Structured Clinical Interview for DSMV (SCID) and clinician-administered measures of mood to determine final study eligibility. This visit will be conducted virtually to limit the number of in-person study visits. At the outset of this visit, all participants will receive verbal and written explanation of the general goals and risks of the study and will virtually sign an informed consent.

The results of the SCID will be used to characterize the study population and to determine whether they meet criteria for any diagnoses that would preclude participation (e.g. psychotic disorders). Their medical history will be reviewed by a study staff member to ensure that patients are diagnostically eligible.

At-home Sleep Recording For 7 days prior to the in-lab study visit, participants will be asked to keep an at-home sleep schedule, consistent with their habitual sleep/wake schedule (e.g., 10:30 PM 6:00 AM). Participants will also consent to refraining from napping, using alcohol and drugs, and limiting caffeine use to one caffeinated beverage before noon on the day of study. These procedures will be confirmed using sleep diary. Sleep diaries will be completed via the REDCap web-based application if participants feel comfortable with an internet-based platform and have consistent Internet access. Paper and pencil versions of sleep diaries will also be available. Study staff will compare across these methods to verify adherence to study guidelines prior to the in-lab study.

In-laboratory Study Protocol Throughout in-laboratory period, participants will be continuously behaviorally monitored by trained staff in a semi-isolated living area, and have contact with only nurses and research. No caffeinated products will be allowed. When not being tested during the study, participants will be permitted to watch television, converse with the study monitors or play games. Physical activity will be kept to a minimum to avoid any effect of exercise on circadian rhythms or sleep. They will not be allowed to leave the study venue.

Day 1 (D1) Participants will arrive at the Clinical Research Center for Sleep (CRCS) in the afternoon of their scheduled overnight, at no later than 1700h. Following their arrival and orientation, participants are accompanied to the MRI for the neuroimaging protocol to acquire data on rested baseline brain activity before sleep deprivation. Following the neuroimaging protocol, participants will return to CRCS and complete mood assessments (HAM-D, PANAS, VAS, POMS).

Night 1 (N1; Sleep deprivation). Sleep will not be permitted from the end of D1 until 1400h on D2 (approximately 30 hours).

Day 2 (D2) Following breakfast at approximately 0700h, all participants will again complete mood assessments. Participants will complete the neuroimaging protocol again between 0900-1200h. Following the neuroimaging protocol, participants will be discharged or allowed to remain in the CRCS for recovery sleep.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 85 years; Current depression as assessed on the SCID;

Stable, normally-timed sleep-wake cycle as determined by interview, 1 week daily sleep log, and defined by:

1. Habitual nocturnal sleep duration between 6h and 9h.
2. Habitual morning awakening between 0600h and 0800h. Able to comprehend English, as all questionnaires are in this language Ability to provide informed consent

Exclusion Criteria:

Shift work, transmeridian travel or irregular sleep/wake routine in past 60 days; A sleep disorder other than insomnia, as determined by history or actigraph; History of bipolar disorder, delirium, dementia, amnestic disorder, schizophrenia and other psychotic disorders as assessed on the SCID; Previous electroconvulsive therapy in the past 6 months; Alcohol or drug abuse in the past year based upon the SCID or urine toxicology screen; A current smoker; Any significant medical or neurological illness that impacts brain function or impedes participation; History of head trauma with significant loss of consciousness; Metallic implants, pacemakers or tattoos, or other contraindications to MRI; Claustrophobic, or intolerant of the scanner environment; Visual or auditory impairment severe enough to compromise task performance as judged by the PI; For women, pregnancy will exclude participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This pilot study is targeting N=10 subjects (10 depressed patients). We will recruit outpatients with current depression from the Philadelphia and University of Pennsylvania community.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
GluCEST imaging metrics | after 24 hours of sleep deprivation
  relative change in glutamate concentration (% baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No